CLINICAL TRIAL: NCT04027153
Title: The Deliver Health Study: A Prospective, Interventional, Randomized Study of Fee for Home ART Delivery in KwaZulu-Natal, South Africa
Brief Title: The Deliver Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ruanne Barnabas, Associate Professor, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00005739; R21MH115770 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-07-19 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: one to one on an individual level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fee Arm (Experimental): Participants in this arm will pay a fee (based on an income sliding scale) to have their medication delivered to their location of choice.
  Interventions: Other: Fee based delivery
- Standard of Care Arm (Active Comparator): Participants in this arm will pick up their medication refill at the local clinic
  Interventions: Other: Fee based delivery

INTERVENTIONS:
Other: Fee based delivery — Testing willingness to pay for services to simplify delivery is innovative as the strategy could increase funds for HIV care making home delivery cost neutral.

SUMMARY:
The investigators hypothesize that routing algorithm based ART delivery will be acceptable, efficient and improve health outcomes, specifically through meeting client needs, retaining HIV-positive persons in care, and achieving high ART resupply and viral suppression. They also hypothesize that a fee for home delivery will improve retention and viral suppression among persons willing to pay a fee for ART delivery. The investigators propose to test ART delivery using routing science and fee for home delivery as strategies that could be scaled-up to sustain lifelong ART.

DETAILED DESCRIPTION:
In KwaZulu-Natal (KZN), South Africa (SA), after an abrupt decline in the 1990s, life expectancy has dramatically rebounded - all driven by the tremendous progress in earlier initiation, once daily, and greater access to ART.23 Efficient ART delivery is key for increasing population coverage and maintaining suppression for life. However, in SA, of the 7.1 million HIV-positive persons, 56% are on ART, and only 45% are virally suppressed (the key indicator of treatment success). Men are less likely to be suppressed than women, due to barriers to care including clinic bottle-necks in ART provision. On a given day, up to 70% of a facility's prescription load is devoted to servicing repeat ART prescriptions. HIV-associated mortality continues to be high, particularly among hard to reach populations who do not regularly visit the clinic on a sufficiently frequent schedule to maintain uninterrupted ART and viral suppression. Over four years, a third of HIV-positive persons in SA are no longer retained in care. Clinically stable HIV-positive persons can safely and effectively receive ART resupply and monitoring in the community. In SA, efforts to deliver medications outside the clinic through the Centralised Chronic Medicines Dispensing and Distribution (CCMDD), led by Project Last Mile (PLM), are focused in urban areas. Data are needed on client preferences for modes of delivery in rural areas, as are innovative, high impact strategies to simplify ART delivery and facilitate life-long ART.

Decentralized ART resupply and monitoring supports successful differentiated service delivery (DSD). Differentiated service delivery (DSD) for HIV (i.e. a client-centered approach that simplifies and adapts services to reflect preferences and expectations of clients while reducing unnecessary burdens on the health system) has the potential to deliver HIV treatment, remove barriers to care, increase retention on ART, and ultimately prevent disability and death at a lower cost. DSD may also have the advantage of de-bulking the clinic allowing providers to focus on clients with medically complex cases. However, there is a fundamental need to match the demand for ART resupply and monitoring with the ART supply, accounting for client preferences for resupply from a local mobile van or at home for convenience and to avoid stigma at the clinic.

The goal of data-driven delivery algorithms is to match ART supply with demand. Amazon.com, the largest internet-based retailer globally, uses routing science extensively and is established in South Africa. Enormous expertise and successful implementation of efficient, low-cost, on-time delivery in diverse settings have been applied by Amazon to get goods to the right person at the right time. Amazon is building their capacity for delivery to rural areas in South Africa, the investigators target geographic location. Since minimal financial resources are available (NDoH pays ZAR 9.36 = USD 0.75 per refill) delivery optimization is essential. The classic computer science Travelling Salesman Problem is used to optimize vehicle routing for delivery through computer algorithms.

Specifically, the investigators propose to adapt vehicle routing algorithms to determine the placement of mobile vans for ART resupply and monitoring in the community. The study area is divided into community clusters of HIV-positive persons who require ART resupply and monitoring. Currently, the study coordinator decides on a weekly basis where the mobile van should be placed, which may not adequately account for multiple cofactors (distance, travel time, client availability). A routing algorithm would efficiently match ART demand with the supply and determine mobile van placement. Importantly, algorithms can use the enrollment GPS location of clients and do not require formal addresses. Routing science guided delivery has the potential to increase efficiency and coverage of ART resupply and monitoring, reduce logistic barriers for clients, and improve the cost efficiency to the health system.

The theoretical basis for proposing ART delivery to increase retention in care and viral suppression is implementation intention i.e. a strategy that automates action control such as planning to collect medication within a given window of availability or having the medication delivered. A fee for the service of home delivery of ART could also increase commitment to care through simplifying ART resupply, addressing logistic barriers (transportation costs, clinic hours), increasing perceived value, and strengthening implementation intentions. To address this separation between intention and action (unsuccessful intenders), cues and plans support engagement in health. Meta-analyses have demonstrated that implementation intentions have medium to large sized effects on behavioral outcomes. Paying a modest fee for home delivery has the potential to increase implementation intention through immediacy and the redundancy of further "conscious intent" (i.e. no additional planning required for clinic collections), simplifying the resupply process. Practically, a fee for home delivery could offset some of the costs of decentralized delivery, making it more appealing to government/investors.

Conceptual model for strengthening ART delivery: Concerns about decentralized ART delivery include how clients would access clinic care, the need for providers to monitor ART, implementation challenges, and concerns about disclosure with home ART delivery. To address these concerns, the investigators are using the evidence integration approach, adapted from Glasgow and colleagues in the investigators current Delivery Optimization for ART (DO ART) Study. The investigators are working with key stakeholders at the department of health, policy makers, clients, and advocates to review evidence and rationale behind decentralized ART delivery and monitoring and assess how to target strategies for scale-up.

Preliminary data: In a series of studies, which demonstrate the investigators capacity to conduct rigorous evaluation of community-based HIV testing and linkage strategies, and utilize study results including costs to contribute to policy, the investigators demonstrated that community-based HIV testing and counseling (HTC) results in >90% knowledge of serostatus and similarly high linkage rates for HIV-positive persons to HIV clinic, which was cost-effective. Results from the investigators work supported the World Health Organization HIV testing guidelines. However, drop-offs in HIV care resulted in only 60% of ART-eligible persons achieving viral suppression (the Linkages Study). Logistic barriers at the clinic such as long wait times, inconvenient hours, and multiple visits are barriers to sustained ART adherence. Preliminary data on spatial analyses: In the Linkages Study the investigators collected GPS data on the location of households and clinics and road map distances. These data demonstrate the investigators ability to collect and utilize geospatial data in statistical analyses.

Significance summary: the investigators hypothesize that routing algorithm based ART delivery will be acceptable, efficient and improve health outcomes, specifically through meeting client needs, retaining HIV-positive persons in care, and achieving high ART resupply and viral suppression. They also hypothesize that a fee for home delivery will improve retention and viral suppression among persons willing to pay a fee for ART delivery. The investigators propose to test ART delivery using routing science and fee for home delivery as strategies that could be scaled-up to sustain lifelong ART.

This proposal is highly innovative and creative in three ways. First, while simplified, decentralized client- centered ART delivery is essential for successful scale-up and lifelong adherence, current strategies do not use routing science methods and are not client-centered; they rely on existing businesses for pick-up points in urban areas. Working closely with the world's largest, successful internet retailer (Amazon.com), the investigators will adapt highly successful delivery algorithms methods to efficiently supply ART in rural settings outside of existing formal facilities utilizing client data on resupply needs, delivery preferences, and availability for pick-up. Second, they will leverage GPS guided delivery in areas without a formal address system, thus increasing overall coverage for decentralized ART delivery. Third, a small fee paid by the client could offset costs of home delivery in a system with an extremely small margin (ZAR 9.36 = USD 0.75 is paid by NDoH for each medication pick-up conducted by CCMDD in the private urban sector). Testing willingness to pay for services to simplify delivery is innovative as the strategy could increase funds for HIV care making home delivery cost neutral.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected and clinically stable
* Eligible for ART according to national guidelines
* Willingness to reside in study community for duration of follow up
* Able and willing to sign the informed consent form
* Willing to pay for medication delivery
* Not known to be pregnant

Exclusion Criteria:

* No separate criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
Number of participants in the Fee arm that paid for delivery | 6 months
  Paying a fee for home delivery of ART demonstrates feasibility and increases the proportion of HIV-positive persons achieving viral suppression, through simplifying resupply and monitoring, and is cost neutral.

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne V Barnaba, MBChB, DPhil, Principal Investigator — University of Washington
Locations (1):
- HSRC Sweetwaters, Sweetwaters, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng AS, Mugwanya KK, Szpiro AA, van Heerden A, Ntinga X, Schaafsma TT, Barnabas RV. Estimating the Effect of COVID-19 Pandemic Restrictions on Self-reported Antiretroviral Therapy Use and Late Refill Visits Among People Living With HIV in Rural South Africa. J Acquir Immune Defic Syndr. 2024 Aug 1;96(4):318-325. doi: 10.1097/QAI.0000000000003431. PMID 38916425
- [Derived] Barnabas RV, Szpiro AA, Ntinga X, Mugambi ML, van Rooyen H, Bruce A, Joseph P, Ngubane T, Krows ML, Schaafsma TT, Zhao T, Tanser F, Baeten JM, Celum C, van Heerden A; Deliver Health Study Team. Fee for home delivery and monitoring of antiretroviral therapy for HIV infection compared with standard clinic-based services in South Africa: a randomised controlled trial. Lancet HIV. 2022 Dec;9(12):e848-e856. doi: 10.1016/S2352-3018(22)00254-5. Epub 2022 Nov 3. PMID 36335976